CLINICAL TRIAL: NCT02732938
Title: PHASE 1B/2 STUDY OF PF-04136309 IN COMBINATION WITH GEMCITABINE AND NAB-PACLITAXEL IN PATIENTS WITH PREVIOUSLY UNTREATED METASTATIC PANCREATIC DUCTAL ADENOCARCINOMA
Brief Title: Ph1b/2 Study of PF-04136309 in Combination With Gem/Nab-P in First-line Metastatic Pancreatic Patients
Acronym: CCR2i
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pfizer made a business-related decision on 04May2017 to terminate study based on change in portfolio prioritization, and is not due to safety or efficacy.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A9421018; 2015-003767-11 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-04-11 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: CCR2i, nab-paclitaxel, Abraxane, gemcitabine, pancreas
MeSH Terms: interventions — PF-04136309; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-04136309 + Nab-p + Gem (Experimental): PF-04136309 oral dosing
  Nab-paclitaxel IV dosing Gemcitabine IV dosing
  Interventions: Drug: PF-04136309; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: PF-04136309 — PF-04136309 oral dosing
Drug: Nab-paclitaxel — Nab-paclitaxel IV dosing
  Other Names: Abraxane
Drug: Gemcitabine — Gemcitabine IV dosing
  Other Names: Gemzar

SUMMARY:
The purpose of this Phase 1b/2 study is to evaluate the safety and tolerability of PF-04136309 in combination with nab-paclitaxel and gemcitabine, characterize the dose-limiting toxicities (DLTs) and overall safety profile of escalated doses of PF-04136309 and the associated schedule, determine the maximum tolerated dose (MTD), and to assess the enhancement of efficacy of PF-04136309 in combination with nab-paclitaxel and gemcitabine versus nab-paclitaxel + gemcitabine + placebo in terms of Progression Free Survival.

DETAILED DESCRIPTION:
The study has 2 parts:

Phase 1b (dose-finding cohorts) will be open label as patients will receive ascending doses of PF-04136309 in combination with nab-paclitaxel + gemcitabine. The observation period for dose-limiting toxicities (DLTs) will be from Day 1 to Day 28. Pharmacokinetic (PK) and pharmacodynamic (PD) properties of PF-04136309 will also be assessed. The criteria for dose escalation will be based on a modified toxicity probability interval (mTPI) method. After evaluating the safety and other results (eg, PK) from patients enrolled in the dose escalation cohorts, a dose level will be selected to be further evaluated as the Recommended Phase 2 Dose (RP2D). A minimum of 6 patients, up to 12 patients, will be treated at this dose level to establish it as the RP2D. To further evaluate safety and pharmacodynamics, the number of patients enrolled during this part of the study (Phase 1b) may be N up to 20. The study will stop if all PF-04136309 doses explored appear to be overly toxic.

Phase 2 randomized double blinded placebo control. Approximately 92 patients will be randomized 1:1 to receive the RP2D of PF-04136309 in combination with nab-paclitaxel + gemcitabine (ARM A; n=46) versus nab-paclitaxel + gemcitabine + placebo (ARM B; n=46). The primary objective will be the enhancement of efficacy in terms of PFS.

Patients will be treated as long as they are clinically benefiting from investigational product without unacceptable toxicity, objective disease progression, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically proven diagnosis of metastatic ductal adenocarcinoma of the pancreas.
2. All patients must provide a baseline tumor sample at registration. If an archival sample is not available, patients must have a metastatic biopsy collected at the screening visit.
3. Patient must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease.
4. Measurable disease as per RECIST v. 1.1.
5. Resolved acute effects of any prior therapy to baseline severity or Grade ≤1 NCI CTCAE.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
7. Age ≥18 years.
8. Adequate Bone Marrow, Renal and liver Functions.

Exclusion Criteria

1. Patients with known symptomatic brain metastases requiring steroids.
2. Prior therapy with modulators of monocyte or TAM function.
3. Participation in other studies involving investigational drug(s) (Phases 1-4) within 4 weeks of registering for the current study and/or during study participation.
4. Diagnosis of any second malignancy within the last 3 years, except for adequately treated basal cell carcinoma, or squamous cell skin carcinoma or in situ cervical carcinoma.
5. Known hypersensitivity to nab-paclitaxel or to gemcitabine or to any of the excipients.
6. Any one of the following currently or in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack; symptomatic pulmonary embolism; congenital long QT syndrome, torsades de points, arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), right bundle branch block and left anterior hemiblock (bifascicular block), ongoing cardiac dysrhythmias of NCI CTCAE Grade >=2, atrial fibrillation of any grade, or QTc interval >470 msec at screening.
7. Concurrent administration of herbal preparations.
8. Use of oral anticoagulants. Use of subcutaneous anti coagulation is allowed. Concurrent use of potent or moderate inhibitors or inducers of CYP3A4 and/or CYP2C8.
9. Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness.
10. History of interstitial lung disease, or slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
11. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior) or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
12. Pregnant female patients; breastfeeding female patients; males patients with partners currently pregnant, male patients able to father children and female patients of childbearing potential who are unwilling or unable to use two (2) highly effective methods of contraception as outlined in this protocol for the duration of the study and for 28 days after last dose of PF-04136309, and for 6 months after last dose of nab-paclitaxel, gemcitabine, or both.
13. Patients who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or patients who are Pfizer employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (17):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center Pharmacy, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Sampson Regional Medical Center, Clinton, North Carolina
  - Southeastern Medical Oncology Center, Clinton, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center, Jacksonville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - MUSC Health East Cooper, Mt. Pleasant, South Carolina
  - MUSC Health North Charleston, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Noel M, O'Reilly EM, Wolpin BM, Ryan DP, Bullock AJ, Britten CD, Linehan DC, Belt BA, Gamelin EC, Ganguly B, Yin D, Joh T, Jacobs IA, Taylor CT, Lowery MA. Phase 1b study of a small molecule antagonist of human chemokine (C-C motif) receptor 2 (PF-04136309) in combination with nab-paclitaxel/gemcitabine in first-line treatment of metastatic pancreatic ductal adenocarcinoma. Invest New Drugs. 2020 Jun;38(3):800-811. doi: 10.1007/s10637-019-00830-3. Epub 2019 Jul 12. PMID 31297636
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9421018&StudyName=Phase%201b%2F2%20Study%20Of%20Pf-04136309%20In%20Combination%20With%20Gemcitabine%20And%20Nab-paclitaxel%20In%20Patients%20With%20Previously%20Untreated%20Metastatic%20Pancreatic%20Ductal%20Adenocarcinoma
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9421018&StudyName=Phase+1b%2F2+Study+Of+Pf-04136309+In+Combination+With+Gemcitabine+And+Nab-paclitaxel+In+Patients+With+Previously+Untreated+Metastatic+Pancreatic+Ductal+Adenocarcinoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 2 part of the study was not conducted due to early termination.
Groups:
- Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine: PF-04136309 (formulated 125 mg tablets) was administered orally at 750 mg twice-daily (BID) for 28-day cycles. Nab-paclitaxel (125 mg/m2) was administered as an intravenous (IV) infusion on Days 1, 8 and 15 followed by 1 week of no treatment in 28-day cycles. Gemcitabine (1000 mg/m2) was administered as an IV infusion immediately after nab-paclitaxel, on Days 1, 8 and 15 followed by 1 week off treatment for 28-day cycles.
- Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine: PF-04136309 (formulated 125 mg tablets) was administered orally at 500 mg BID for 28-day cycles. Nab-paclitaxel (125 mg/m2) was administered as an IV infusion on Days 1, 8 and 15 followed by 1 week of no treatment in 28-day cycles. Gemcitabine (1000 mg/m2) was administered as an IV infusion immediately after nab-paclitaxel, on Days 1, 8 and 15 followed by 1 week off treatment for 28-day cycles.
- Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine: In Phase 2 part of the study which was not conducted due to early termination, participants were to be randomized with a 1:1 to receive either PF-04136309 or placebo in combination with nab-paclitaxel + gemcitabine. The dose of PF-04136309 was to be the recommended Phase 2 dose (RP2D) determined in the Phase 1b part of the study.
Period: Overall Study
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Started | 4 | 18 | 0
Received Treatment | 4 | 17 | 0
Completed | 0 | 0 | 0
Not Completed | 4 | 18 | 0
Not completed — Death | 0 | 11 | 0
Not completed — Randomized but did not receive treatment | 0 | 1 | 0
Not completed — Refused further follow-up | 1 | 0 | 0
Not completed — Study terminated by sponsor | 3 | 6 | 0

BASELINE CHARACTERISTICS:
Population: All Phase 1b enrolled participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine | Total
Number analyzed (Participants) | 4 | 17 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 10 | 12
  >=65 years | 2 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.2) | 61.9 (8.9) | 61.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 0 | 11 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 15 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) [Phase 1b]
Description: DLT: Any of the following events occurred in the first treatment cycle and was attributed to the combination of PF-04136309 with nab-paclitaxel and gemcitabine where relationship with the combination could not be ruled out. Hematologic: Grade (Gr) 4 neutropenia lasting more than (>)5 days; febrile neutropenia; Gr≥3 neutropenic infection; Gr≥3 thrombocytopenia with Gr≥2 bleeding; Gr4 thrombocytopenia. Non-Hematologic: Gr3 toxicities (except: nausea and vomiting responding to prophylaxis and/or treatment and lasting less than (<)7 days from each chemotherapy infusion period; diarrhea responding to treatment and lasting <7 days; Gr3 QTc prolongation [QTc >500 milliseconds] [a DLT only if persisting after correction of any reversible causes]; Gr3 aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) increase lasting less than or equal to (≤)7 days); all Gr4 toxicities; delay of >2 weeks in receiving the next scheduled cycle due to persisting treatment-related toxicities.
Time Frame: Day 1 to Day 28
Population: All Phase 1b enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 17
Participants | 1 | 3

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) [Phase 1b]
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment.
Time Frame: 1 year
Population: All Phase 1b enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 17
Participants
  Treatment-emergent AE (all causality) | 4 | 17
  Treatment-emergent AE (PF-04136309 related) | 3 | 16
  Treatment-emergent SAE (all causality) | 3 | 11
  Treatment-emergent SAE (PF-04136309 related) | 2 | 4

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) by Severity [Phase 1b]
Description: Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment. AEs were graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03: Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: 1 year
Population: All Phase 1b enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 17
Participants
  Grade 1 | 0 | 0
  Grade 2 | 0 | 1
  Grade 3 | 4 | 12
  Grade 4 | 0 | 3
  Grade 5 | 0 | 1

4. Primary Outcome: Number of Participants With Hematology Laboratory Abnormalities by Maximum National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) Grade [Phase 1b]
Description: Following parameters were analyzed for hematology laboratory test: hemoglobin, hematocrit, red blood cell (RBC) count, mean corpuscular volume (MCV); mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), platelet count, white blood cell (WBC) count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes. Laboratory abnormalities were graded per NCI CTCAE version 4.03 and those with at least 1 participant are presented here.
Time Frame: 1 year
Population: All Phase 1b enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 17
Participants
  Anemia, Grade 1 | 1 | 5
  Anemia, Grade 2 | 3 | 8
  Anemia, Grade 3 | 0 | 4
  Lymphocyte count increased, Grade 2 | 0 | 1
  Lymphopenia, Grade 1 | 1 | 3
  Lymphopenia, Grade 2 | 2 | 3
  Lymphopenia, Grade 3 | 1 | 8
  Neutrophils (absolute), Grade 1 | 0 | 1
  Neutrophils (absolute), Grade 2 | 0 | 5
  Neutrophils (absolute), Grade 3 | 3 | 2
  Neutrophils (absolute), Grade 4 | 0 | 1
  Platelets, Grade 1 | 3 | 10
  Platelets, Grade 2 | 1 | 2
  WBC, Grade 1 | 0 | 2
  WBC, Grade 2 | 0 | 5
  WBC, Grade 3 | 3 | 2
  WBC, Grade 4 | 0 | 1

5. Primary Outcome: Number of Participants With Chemistries Laboratory Abnormalities by Maximum NCI CTCAE Grade [Phase 1b]
Description: Following parameters were analyzed for chemistry laboratory test: blood urea nitrogen (BUN), creatinine, glucose (fasting), calcium, sodium, potassium, chloride, total bicarbonate, AST, ALT, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, Magnesium, phosphorous or phosphate. For potential Hy's Law cases, in addition to repeating AST and ALT, laboratory tests should have included albumin, creatine kinase, total bilirubin, direct and indirect bilirubin, gamma-glutamyl transferase (GGT), prothrombin time / international normalized ratio (PT/INR), alkaline phosphatase, total bile acids, and acetaminophen drug and/or protein adduct levels. Laboratory abnormalities were graded per NCI CTCAE version 4.03 and those with at least 1 participant are presented here.
Time Frame: 1 year
Population: All Phase 1b enrolled participants who received at least 1 dose of study treatment. GGT was an additional test for potential Hy's law. Only 1 participant in the PF-04136309 500 mg BID + Nab-paclitaxel + Gemcitabine treatment group was tested for GGT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 17
Participants
  ALT, Grade 1 | 1 | 8
  ALT, Grade 2 | 2 | 3
  ALT, Grade 3 | 1 | 4
  ALT, Grade 4 | 0 | 1
  Alkaline phosphatase, Grade 1 | 2 | 7
  Alkaline phosphatase, Grade 2 | 1 | 5
  Alkaline phosphatase, Grade 3 | 0 | 2
  AST, Grade 1 | 2 | 8
  AST, Grade 2 | 1 | 1
  AST, Grade 3 | 1 | 5
  Bilirubin (total), Grade 1 | 0 | 1
  Bilirubin (total), Grade 2 | 0 | 3
  Bilirubin (total), Grade 3 | 0 | 2
  Creatinine, Grade 1 | 4 | 9
  Creatinine, Grade 2 | 0 | 2
  GGT, Grade 1: number analyzed (Participants) | 0 | 1
  GGT, Grade 1 |  | 1
  Hyperglycemia, Grade 1 | 2 | 6
  Hyperglycemia, Grade 2 | 2 | 6
  Hyperglycemia, Grade 3 | 0 | 5
  Hyperkalemia, Grade 1 | 0 | 2
  Hypermagnesemia, Grade 1 | 0 | 1
  Hypoalbuminemia, Grade 1 | 0 | 8
  Hypoalbuminemia, Grade 2 | 1 | 6
  Hypocalcemia, Grade 1 | 2 | 6
  Hypocalcemia, Grade 2 | 0 | 2
  Hypoglycemia, Grade 2 | 0 | 1
  Hypokalemia, Grade 1 | 1 | 3
  Hypokalemia, Grade 3 | 0 | 1
  Hypomagnesemia, Grade 1 | 1 | 5
  Hyponatremia, Grade 1 | 0 | 7
  Hyponatremia, Grade 3 | 0 | 3
  Hypophosphatemia, Grade 2 | 0 | 3
  Hypophosphatemia, Grade 3 | 0 | 1

6. Primary Outcome: Number of Participants With Urinalysis Laboratory Abnormalities by Maximum NCI CTCAE Grade [Phase 1b]
Description: Following parameters were analyzed for urinalysis laboratory test: pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy (only if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase), urine dipstick for urine protein (if positive collected 24 hour and microscopic [reflex testing]), urine dipstick for urine blood (if positive collected a microscopic [reflex testing]). Laboratory abnormalities were graded per NCI CTCAE version 4.03 and those with at least 1 participant are presented here.
Time Frame: 1 year
Population: All Phase 1b participants who received at least 1 dose of study treatment and had at least 1 post-dose urinalysis laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 16
Participants | 1 | 0

7. Primary Outcome: Progression Free Survival (PFS) [Phase 2]
Description: PFS was defined as the time from randomization to first documentation of objective tumor progression or to death due to any cause, whichever occurred first.
Time Frame: 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

8. Secondary Outcome: PF-04136309 Maximum Observed Plasma Concentration (Cmax) for Cycle 1 Day 15 in the 750 mg BID Group [Phase 1b]
Description: Cmax of PF-04136309 was observed directly from data. This outcome measure reports individual values for the participants in the Phase 1b PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine treatment group as summary statistics were not generated when fewer than 3 participants had reportable data.
Time Frame: Cycle 1 Day 15 pre-dose (within 30 minutes), and 0.5, 1, 2, 3, 4, and 6 hours after the morning dose; Cycle 1 Day 16 pre-dose (within 30 minutes; as the 12-hour sample for evening dose on Day 15)
Population: "Number of participants analyzed" represents all Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Cmax data; "Number analyzed" represents the number of such participants for each category.
Measure: Number; unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 2
nanograms per milliliter (ng/mL)
  Individual value for Participant 1: number analyzed (Participants) | 1
  Individual value for Participant 1 | 3390
  Individual value for Participant 2: number analyzed (Participants) | 1
  Individual value for Participant 2 | 2950

9. Secondary Outcome: PF-04136309 Maximum Observed Plasma Concentration (Cmax) for Cycle 1 Day 15 in the 500 mg BID Group [Phase 1b]
Description: Cmax of PF-04136309 was observed directly from data. This outcome measure reports summary statistics for the participants in the Phase 1b PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine treatment group. Arithmetic coefficient of variation (CV) was the intended method of dispersion for reporting but system only has geometric CV option, hence geometric CV data were reported for this parameter.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 13
ng/mL | 1276 (52)

10. Secondary Outcome: PF-04136309 Time to Reach Maximum Observed Plasma Concentration (Tmax) for Cycle 1 Day 15 in the 750 mg BID Group [Phase 1b]
Description: Tmax of PF-04136309 was observed directly from data as time of first occurrence. This outcome measure reports individual values for the participants in the Phase 1b PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine treatment group as summary statistics were not generated when fewer than 3 participants had reportable data.
Time Frame: as for outcome 8
Population: "Number of participants analyzed" represents all Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Tmax data; "Number analyzed" represents the number of such participants for each category.
Measure: Number; unit: hours (hr)
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 2
hours (hr)
  Individual value for Participant 1: number analyzed (Participants) | 1
  Individual value for Participant 1 | 1.00
  Individual value for Participant 2: number analyzed (Participants) | 1
  Individual value for Participant 2 | 3.02

11. Secondary Outcome: PF-04136309 Time to Reach Maximum Observed Plasma Concentration (Tmax) for Cycle 1 Day 15 in the 500 mg BID Group [Phase 1b]
Description: Tmax of PF-04136309 was observed directly from data as time of first occurrence. This outcome measure reports summary statistics for the participants in the Phase 1b PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine treatment group.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Tmax data.
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 13
hours (hr) | 1.42 [0.500 to 5.95]

12. Secondary Outcome: PF-04136309 Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Cycle 1 Day 15 in the 750 mg BID Group [Phase 1b]
Description: The dosing interval was 12 hours for PF-04136309 BID dosing. AUCtau was determined by linear/log trapezoidal method. This outcome measure reports individual values for the participants in the Phase 1b PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine treatment group as summary statistics were not generated when fewer than 3 participants had reportable data.
Time Frame: as for outcome 8
Population: "Number of participants analyzed" represents all Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had AUCtau data; "Number analyzed" represents the number of such participants for each category.
Measure: Number; unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 2
nanogram*hour/milliliter (ng*hr/mL)
  Individual value for Participant 1: number analyzed (Participants) | 1
  Individual value for Participant 1 | 15700
  Individual value for Participant 2: number analyzed (Participants) | 1
  Individual value for Participant 2 | 10600

13. Secondary Outcome: PF-04136309 Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Cycle 1 Day 15 in the 500 mg BID Group [Phase 1b]
Description: The dosing interval was 12 hours for PF-04136309 BID dosing. AUCtau was determined by linear/log trapezoidal method. This outcome measure reports summary statistics for the participants in the Phase 1b PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine treatment group. Arithmetic CV was the intended method of dispersion for reporting but system only has geometric CV option, hence geometric CV data were reported for this parameter.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had AUCtau data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 13
ng*hr/mL | 5873 (36)

14. Secondary Outcome: PF-04136309 Minimum Observed Plasma Concentration (Cmin) for Cycle 1 Day 15 in the 750 mg BID Group [Phase 1b]
Description: Cmin of PF-04136309 was observed directly from data. This outcome measure reports individual values for the participants in the Phase 1b PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine treatment group as summary statistics were not generated when fewer than 3 participants had reportable data.
Time Frame: as for outcome 8
Population: "Number of participants analyzed" represents all Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Cmin data; "Number analyzed" represents the number of such participants for each category.
Measure: Number; unit: ng/mL
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 2
ng/mL
  Individual value for Participant 1: number analyzed (Participants) | 1
  Individual value for Participant 1 | 436
  Individual value for Participant 2: number analyzed (Participants) | 1
  Individual value for Participant 2 | 0

15. Secondary Outcome: PF-04136309 Minimum Observed Plasma Concentration (Cmin) for Cycle 1 Day 15 in the 500 mg BID Group [Phase 1b]
Description: Cmin of PF-04136309 was observed directly from data. This outcome measure reports summary statistics for the participants in the Phase 1b PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine treatment group.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Cmin data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 13
ng/mL | 72.34 (NA) — NA for geometric coefficient of variation as there were participants with a zero value (ie, Cmin below the limit of quantification).

16. Secondary Outcome: PF-04136309 Apparent Oral Clearance (CL/F) for Cycle 1 Day 15 in the 750 mg BID Group [Phase 1b]
Description: CL/F was determined by Dose/AUCtau. AUCtau is the area under the curve from time 0 to end of dosing interval. This outcome measure reports individual values for the participants in the Phase 1b PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine treatment group as summary statistics were not generated when fewer than 3 participants had reportable data.
Time Frame: as for outcome 8
Population: "Number of participants analyzed" represents all Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had CL/F data; "Number analyzed" represents the number of such participants for each category.
Measure: Number; unit: Liters per hour (L/hr)
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 2
Liters per hour (L/hr)
  Individual value for Participant 1: number analyzed (Participants) | 1
  Individual value for Participant 1 | 47.8
  Individual value for Participant 2: number analyzed (Participants) | 1
  Individual value for Participant 2 | 70.5

17. Secondary Outcome: PF-04136309 Apparent Oral Clearance (CL/F) for Cycle 1 Day 15 in the 500 mg BID Group [Phase 1b]
Description: CL/F was determined by Dose/AUCtau. AUCtau is the area under the curve from time 0 to end of dosing interval. This outcome measure reports summary statistics for the participants in the Phase 1b PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine treatment group. Arithmetic CV was the intended method of dispersion for reporting but system only has geometric CV option, hence geometric CV data were reported for this parameter.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had CL/F data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 13
Liters per hour (L/hr) | 85.09 (36)

18. Secondary Outcome: PF-04136309 Plasma Decay Half-Life (t1/2) for Cycle 1 Day 15 [Phase 1b]
Description: t1/2 was determined by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had t1/2 data.
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 1 | 10
hours (hr) | 1.18 (NA) — NA for standard deviation as only 1 participant had data for t1/2. | 3.41 (0.996)

19. Secondary Outcome: PF-04136309 Apparent Volume of Distribution (Vz/F) for Cycle 1 Day 15 [Phase 1b]
Description: Vz/F was determined by Dose/(AUCtau×kel). AUCtau is the area under the curve from time 0 to end of dosing interval and kel is the terminal phase rate constant.
Time Frame: as for outcome 8
Population: All Phase 1b participants who received planned treatments on Cycle 1 Day 15 and had Vz/F data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 1 | 10
Liters (L) | 120 (NA) — NA for geometric coefficient of variation as only 1 participant had data for Vz/F. | 398.3 (NA) — NA for geometric coefficient of variation as there were missing values for Vz/F.

20. Secondary Outcome: Ex Vivo Inhibition of Chemokine Ligand 2 (CCL2)-Induced Extracellular Signal Regulated Kinase (ERK) Phosphorylation in the Peripheral Blood [Phase 1b]
Description: A drop in the CCL2-induced ERK kinase phosphorylation (pERK) biomarker level indicates target engagement (TE).
Time Frame: Cycle 1 Day 1 pre-dose, 2 and 6 hours post-dose, and 12 hours (pre-second BID dose-optional collection); Cycle 1 Days 2, 3 and 4 pre-dose
Population: No data to report for this outcome measure as only individual plots were planned and generated to show the trend of biomarker level in each participant. Summary statistics were not planned and hence not generated.
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 0 | 0

21. Other Pre Specified Outcome: Objective Response Rate (ORR) [Phase 1b]
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) according to the Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1, relative to all randomized participants who had baseline measurable disease. Confirmed responses were those that persisted on repeat imaging study ≥4 weeks after initial documentation of response.
Time Frame: 1 year
Population: All the Phase 1b treated participants with measurable disease baseline assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
Number analyzed (Participants) | 4 | 17
Percentage of Participants | 0 [0 to 60.2] | 29.4 [10.3 to 56.0]

22. Secondary Outcome: Number of Participants With Overall Survival (OS) [Phase 2]
Description: OS was defined as the time from date of randomization to date of death due to any cause. For participants not expiring, their survival times were to be censored at the last date they were known to be alive. Participants lacking data beyond the day of randomization were to have their survival times censored at the date of randomization with duration of 1 day.
Time Frame: Up to approximately 13.5 months
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) [Phase 2]
Description: An AE was any untoward medical occurrence in a participant administered a product or medical device without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study treatment.
Time Frame: Up to approximately 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

24. Secondary Outcome: Number of Participants With Laboratory Abnormalities by Severity [Phase 2]
Description: Hematology, chemistry, and urinalysis laboratory parameters were to be analyzed and graded by NCI CTCAE version 4.03.
Time Frame: Up to approximately 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

25. Secondary Outcome: Objective Response Rate (ORR) [Phase 2]
Description: as for outcome 21
Time Frame: Up to approximately 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

26. Secondary Outcome: Duration of Objective Response (DR) [Phase 2]
Description: DR was defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first. DR data were to be censored on the day following the date of the last on treatment (including 28 day follow-up period after last dose) tumor assessment documenting absence of progressive disease for participants who did not have objective tumor progression and who did not die due to any cause while on treatment or who were given anti-tumor treatment other than the study treatment prior to observing objective tumor progression. Participants who achieved a PR and then a CR were to have times calculated using the date of the PR as the first day. DR was only to be calculated for the subgroup of participants with objective response.
Time Frame: Up to approximately 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

27. Secondary Outcome: Time to Progression (TTP) With the Double Combination PF-04136309 and Gemcitabine (Maintenance Therapy) After Interruption of Nab-paclitaxel [Phase 2]
Description: This type of TTP was defined as the time from interruption of nab-paclitaxel to the first documentation of objective tumor progression. This TTP was to be only calculated for the subgroup of participants who were treated with the maintenance therapy.
Time Frame: Up to approximately 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

28. Secondary Outcome: Trough PF-04136309 Concentrations [Phase 2]
Description: The minimum plasma concentration of PF-04136309.
Time Frame: Cycle 1 Day 1 pre-dose, Cycle 1 Days 2, 8 and 15 pre-dose; Day 1 of Cycle 2 and subsequent cycles pre-dose, and EOT visit
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

29. Secondary Outcome: Change From Baseline in Pharmacodynamic (PD) Markers in Metastatic Tumors and Bone Marrow [Phase 2]
Description: Collections of core needle biopsy (CNB) from a metastatic site or fine-needle aspirate (FNA) from the primary tumor tissue were optional but at least 12 paired biopsies would have to be available and fully assessable in each treatment arm to allow the comparison.
Time Frame: Baseline, Cycle 1 Day 28 or Cycle 2 Day 28; EOT visit (optional) for CNB
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

30. Secondary Outcome: Number of Participants With Peripheral Neurological Adverse Events [Phase 2]
Description: To evaluate the improvement of peripheral neurotoxicity induced by nab-paclitaxel by the addition of PF-04136309 to the combination therapy of nab-paclitaxel plus gemcitabine.
Time Frame: Up to approximately 1 year
Population: No data to report as Phase 2 part was not conducted.
Arm/Group | Phase 2: PF-04136309 or Placebo + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from baseline through 28 days after last dose of study treatment (up to approximately 1 year).
Description: Survival status was collected every 3 months after treatment discontinuation. A total of 11 deaths were reported, 1 of which was within AE reporting time frame (within 28 days after last dose of study treatment) and 10 of which were after AE reporting time frame (after 28 days following last dose of study treatment).
Arm/Group | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/4 | 11/17
Serious Adverse Events (participants affected / at risk) | 3/4 | 11/17
Other Adverse Events (participants affected / at risk) | 4/4 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine (N=4) | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine (N=17)
Episcleritis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Biliary sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: PF-04136309 750 mg BID +Nab-paclitaxel +Gemcitabine (N=4) | Phase 1b: PF-04136309 500 mg BID +Nab-paclitaxel +Gemcitabine (N=17)
Anaemia (Blood and lymphatic system disorders) | 2 | 11
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 3 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 14
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pancreatic failure (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 7
Asthenia (General disorders) | 0 | 3
Chest discomfort (General disorders) | 0 | 3
Chills (General disorders) | 2 | 4
Device related thrombosis (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Early satiety (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 13
Malaise (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 8
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 2 | 10
Suprapubic pain (General disorders) | 1 | 0
Xerosis (General disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2
Alanine aminotransferase (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 7
Aspartate aminotransferase (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 6
Blood albumin (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 7
Blood bilirubin increased (Investigations) | 0 | 4
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Immunoglobulins decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 4
Monocyte count increased (Investigations) | 0 | 1
Neutrophil count (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 0 | 3
Weight decreased (Investigations) | 1 | 9
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 4
White blood cells urine positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 0 | 4
Dysaesthesia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 2
Fine motor skill dysfunction (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 5
Mental impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 9
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 3
Depression (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 8
Chromaturia (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 0 | 2
Infarction (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated prematurely based on the company's change in prioritization for the portfolio and was not due to any safety concerns or regulatory interactions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT02732938/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02732938/SAP_001.pdf